CLINICAL TRIAL: NCT00418535
Title: A Phase II Study of Concurrent Chemoradiation Followed by VIPD (Etoposide/Ifosfamide/Cisplatin/Dexamethasone) in Stage I, II Nasal NK/T-cell Lymphoma
Brief Title: Clinical Study of Chemoradiation Followed by VIPD in Nasal Natural Killer (NK)/T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korea University Anam Hospital (Other); Asan Medical Center (Other); Gyeongsang National University Hospital (Other)
Responsible Party: CISL (Consortium to Improve Lymphoma Survival), CISL (Consortium to Improve Lymphoma Survival)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-10-08
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2007-01

CONDITIONS: Lymphoma, T-Cell
Keywords: Lymphoma, NK/T-Cell
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma

INTERVENTIONS:
Drug: Concurrent Radiotherapy (RT)/cisplatin, VIPD

SUMMARY:
Nasal NK/T-cell lymphoma is a peculiar clinico-pathologic subtype of non-Hodgkin's lymphoma (NHL). Although most patients present with stage I/II, only 30-60% of the patients remain disease-free. The efficacy of the conventional anthracycline-based chemotherapy (cyclophosphamide, doxorubicin, vincristine, prednisone [CHOPP]) has been unsatisfactory.

The optimal treatment of localized NK/T-cell lymphoma has not been defined yet. The optimal dose, sequence, and multi-modality treatment with involved field radiotherapy still need to be refined. This trial is to evaluate the efficacy of concurrent chemoradiotherapy with cisplatin followed by VIPD (etoposide, ifosfamide, cisplatin, dexamethasone) in localized NK/T-cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed NK/T-cell lymphoma
* Localized (Ann Arbor stage I/II) disease
* At least one measurable lesion
* Age > 18
* ECOG performance status 0 - 2
* Expected life span of at least 12 weeks
* Normal marrow function (hemoglobin ≥ 9.0 g/dL; absolute neutrophil count ≥ 1,500/mm3; platelet count ≥ 100,000/mm3)
* Normal liver function (total bilirubin < 2x upper limit of normal [ULN], transaminase < 3x ULN)
* Normal renal function (serum creatinine ≤ 1.5 mg/dL, creatinine clearance ≥ 50 mL/min)
* Written informed consent

Exclusion Criteria:

* Other malignancies except for treated non-melanoma skin cancers and cervical cancer in situ
* Serious medical illnesses (congestive heart failure, angina, respiratory failure, and renal failure)
* Acute or active infection requiring intravenous (IV) antibiotics
* Pregnant, lactating women
* Previous history of chemotherapy or radiotherapy
* Concomitant medication that may influence the study drugs
* Allergic reaction to study drugs
* Grade 2 or greater peripheral neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-04; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea